CLINICAL TRIAL: NCT05792761
Title: A Study on Antiviral Treatment of Chronic Hepatitis B in Children (Sprout Project)
Brief Title: A Study on Antiviral Treatment of Chronic Hepatitis B in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fang Wang (Other)
Responsible Party: Sponsor-Investigator, Fang Wang, Chief physician, Shenzhen Third People's Hospital
Organization: Shenzhen Third People's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sprout project
Record Dates: First submitted 2023-02-23; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Chronic HBV Infection
MeSH Terms: interventions — entecavir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- treatment-naïve children with hepatitis B (Experimental)
  Interventions: Drug: Peginterferon alfa-2b combined and ETV
- previously treated children with hepatitis B (Experimental)
  Interventions: Drug: Peginterferon alfa-2b combined and ETV
- chronic HBV carrying children with normal ALT (Experimental)
  Interventions: Drug: Peginterferon alfa-2b combined and ETV

INTERVENTIONS:
Drug: Peginterferon alfa-2b combined and ETV — Child patients are assigned to one of the 3 treatment regimens according to their illness state and treatment desire of their parents/guardians, and the number of patients in each group is expected to limited to 300.
  1. NA monotherapy group : received entecavir (ETV) for 96 weeks.
  2. Combination therapy group: received peginterferon alfa-2b combined with ETV for 96 weeks.
  3. Pulse therapy group :received peginterferon alfa-2b pulse treatment combined with ETV for 144 weeks.

SUMMARY:
There are nearly 2 million HBsAg-positive children who are in urgent need of professional diagnosis and treatment in China. Chronic hepatitis B (CHB) is the leading cause of childhood liver disease. After infected with HBV virus, some children will develop disease progression, and some even develop cirrhosis and/or liver cancer. In pediatric liver cancer cases, up to 34% ~ 95% are caused by HBV infection.

Although two major classes of drugs have been approved for the treatment of chronic hepatitis B in adults, and there are multiple guidelines worldwide for the management of HBV infection in adults, there is lack of guidelines specifically for the management of children with HBV infection. In addition, the treatment of chronic hepatitis B in children faced great difficulties due to the lack of evidence-based medical evidence for antiviral treatment of chronic hepatitis B in children and fewer drugs approved for anti-HBV treatment in children. The timing of treatment, medications, and clinical management strategies are all controversial.

This study ( Sprout project)，is a multicenter, prospective, cohort study in China, aiming to explore and optimize the antiviral treatment regimen for children with HBV infection, to provide evidence-based medical for antiviral treatment, and to provide basis evidence for the standardized management of children infection with HBV in China. The study is expected to enroll 1900 pediatric patients with HBV infection, and patient will received one of the three following treatment Strategies: nucleoside monotherapy, peginterferon α- combined with nucleoside therapy, or peginterferon α-pulse therapy combined with nucleoside therapy, according to their illness state and desire, and the safety and efficacy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1.Inclusion criteria for treatment-naïve children with hepatitis B:

1. Aged 3 to 18 (included 3 years old, but exclude 18 years old);
2. HBV DNA positive (higher than the lower detection limit or >20 IU/ml. Roche reagent is recommended).
3. HBsAg positive (higher than lower detection limit or >0.05 IU/ml. Roche reagent is recommended).
4. ALT flares between 1 to10 ULN at least twice a year. If the last examination result is higher than 5ULN, the investigator shall comprehensively judge whether the child patient is suitable to participate in this study.
5. The guardian should understand and sign the informed consent form (if parents is the legal guardians, they both must sign the informed consent form). Children older than 8 years (included) also must sign the informed consent form. The consent comment of child patient under the age of 8 should also be clearly recorded.

2.Inclusion criteria for NA-treated children with hepatitis B:

1. Aged 3 to 18 (included 3 years old, but exclude 18 years old);
2. Previously received NA treatment for ≥ 1 year.
3. HBsAg positive (higher than lower detection limit or >0.05 IU/ml. Roche reagent is recommended).
4. The guardian should understand and sign the informed consent form (if parents is the legal guardians, they both must sign the informed consent form). Children older than 8 years (included) also must sign the informed consent form. The consent comment of child patient under the age of 8 should also be clearly recorded.

3.Inclusion criteria for chronic HBV carrying children with normal ALT:

1. Aged 3 to 18 (included 3 years old, but exclude 18 years old);
2. HBV DNA positive (higher than lower detection limit or >20 IU/ml. Roche reagent is recommended).
3. HBsAg positive (higher than lower detection limit or >0.05 IU/ml. Roche reagent is recommended).
4. Serum ALT and AST remain persistently normal (2 consecutive follow-up visits within half a year, with an interval of at least 3 months)
5. TThe guardian should understand and sign the informed consent form (if parents is the legal guardians, they both must sign the informed consent form). Children older than 8 years (included) also must sign the informed consent form. The consent comment of child patient under the age of 8 should also be clearly recorded.

Exclusion Criteria:

1. Co-infected with HAV, HCV, HDV, HEV or HIV.
2. Patients with contraindications to peginterferon alfa-2b, including but not limit to :

   1. Hepatitis B cirrhosis decompensated stage.
   2. Child patient with autoimmune liver disease, metabolic liver disease or alcoholic liver disease; malignant tumor, decompensated liver disease, or organ transplantation.
   3. Child patient with severe neurological or mental disorders.
   4. Child patient with severe hyperthyroidism or other autoimmune disorders.
   5. Child patient with diabetes under poorly controlled.
   6. Child patient with retinal or fundus lesions.
   7. Child patient with severe heart disease, coronary heart disease or cerebrovascular disease.
   8. Child patient with poorly controlled epilepsy.
3. Child patient with severe renal dysfunction, e.g. creatinine > 1.5 ULN.
4. Child patient who in the opinion of the investigator is unsuitable for enrollment.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1900 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate. | 24 weeks after completing treatment.
  Defined as the proportion of child patients with HBsAg < 0.05 IU / mL (or below the lower detection limit) 24 weeks after completing treatment, HBeAg negative, HBV DNA undetectable, and normalization of liver biochemical indexes (ALT and AST).

SECONDARY OUTCOMES:
Proportion of patients with HBV-DNA negative in those with HBV-DNA positive at baseline. | 24 weeks after treatment completion
  Defined as HBV-DNA below the lower detection limit, or< 20 IU/mL.
HBeAg seroconversion rate in HBeAg positive children. | 24 weeks after treatment completion.
  Defined as HBeAg negative and anti-HBe positive.
HBsAg seroconversion rate. | 24 weeks after treatment completion.
  Defined as HBsAg < 0.05 IU/mL and anti-HBe positive.
ALT normalization rate. | 48 weeks and 96 weeks after starting treatment
Decrease of HBV-DNA compared to baseline. | 24 weeks after treatment completion.
Decrease of HBeAg compared to baseline. | 24 weeks after treatment completion.
Decrease of HBsAg compared to baseline. | 24 weeks after treatment completion.
The incidence of adverse reactions. | 24weeks ,48 weeks and 96 weeks after starting treatment
  Including fever, influenza-like symptoms, decreased hemogram, jaundice ALT> 400U/L, abnormal renal function, abnormal thyroid function, abnormal blood phosphorus and blood calcium during treatment (lower or higher than the normal value).
The effects on height | 24weeks ,48 weeks and 96 weeks after starting treatment
The effects on weight | 24weeks ,48 weeks and 96 weeks after starting treatment
The effects on bone age. | 24weeks ,48 weeks and 96 weeks after starting treatment

CONTACTS AND LOCATIONS:
Overall Officials: Qing He, Principal Investigator — Shenzhen Third People's Hospital; Hongfei Zhang, Principal Investigator — Beijing Tsinghua Changgeng Hospital; Fang Wang, Study Chair — Shenzhen Third People's Hospital
Locations (1):
- Shenzhen Third People Hospital, Shenzhen, China

IPD SHARING:
Plan to Share IPD: No